CLINICAL TRIAL: NCT06249594
Title: Real-World Treatment Patterns, Clinical Outcomes of a Novel Method in Targeted Sensory Re-innervation in Hand Amputation by Using and Reactivation of Existing Nerves to Treat and Prevent Phantom Pain A Retrospective, Non-interventional, Multinational, Multi-center Retrospective Data Analysis to Describe the Treatment Patterns and Clinical Outcomes in a Novel Method in Targeted Sensory Reinnervation in Patients With Hand Amputation by Using and Reactivation of Existing Nerves to Treat and Prevent Phantom Pain.
Brief Title: Targeted Sensory Reinnervation (TSR) in Hand Amputation
Status: Completed | Type: Observational
Sponsor: Brixsana Private Clinic - Centro di Chirurgia Plastica, Estetica ed Ricostruttiva con Chirurgia dell (Other)
Collaborators: AUVA Hospital Klagenfurt/Austria (Unknown); Ludwig Boltzmann Institute for Traumatology - The research center in cooperation with AUVA (Other Government); CCSRM - Clinical Center for Studies in Regenerative Medicine (Unknown)
Responsible Party: Sponsor
Other Study IDs: TSR in Hand Amputation
Record Dates: First submitted 2024-01-23; First posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-01

CONDITIONS: Targeted Sensory Reinervation; Amputation; Phantom Pain
Keywords: Nerves; Reinervation; amputation hand; phantom pain; prevention; novel methode
MeSH Terms: conditions — Phantom Limb

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: targeted sensory reinervation — targeted sensory reinnervation (TSR) in hand amputation by using and reactivation of existing nerves to treat and prevent phantom pain

SUMMARY:
If a person has to have a part of their body amputated, in this case their hand, the patient then lacks information about the missing limb, which in many cases leads to pain that severely restricts their quality of life and participation in everyday life.

This is usually phantom and/or neuroma pain. Phantom pain is usually caused by many different mechanisms and occurs in 80-90% of patients.

Pain caused by terminal neuromas affects 13-32% of amputees and manifests itself as residual limb pain.

A neuroma itself is a benign lump that can develop at the site of the defect after a nerve has been severed (neurectomy).

In some cases the impairment is so severe that prosthetic tolerance, functional independence and quality of life can be severely affected.

Numerous treatment options for these types of pain are far from satisfactory for many patients and remain a major challenge for both the clinician and the person affected.

It is often no longer possible for the patients to pursue a profession or hobby due to the pain as well as due to the pain medication required and its possible side effects.

Surgical intervention can therefore be considered for patients who do not (or no longer) respond to conservative pain treatment.

In recent years, many surgical approaches have been introduced to treat or prevent post-amputee pain.

One of these methods can make it possible to create an authentic feeling of the missing limb and thus reduce or eliminate phantom pain by means of targeted sensory reinnervation (TSR) of the lost body part.

Sensory reinnervation means that a nerve which enables a (sensory) perception associated with a sense is "redirected" to a new area of the body and can therefore fulfil at least part of its task again.

In this case, an authentic feeling of the lost body part.

The aim of this retrospective data-analysis is to evaluate data from patients with hand amputation (planned surgery or caused by accident/infection..) who have undergone TSR surgery to treat or prevent phantom and neuro-pain with regard to different parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patients with amputations of the hand
* Patient with programmed hand amputation
* Patients with treatment-resistant pain
* Patients with treatment-resistant phantom- and neuroma pain
* Patients with performed TSR Surgery
* Aged at least 18 years
* Patient must be alive at the time of medical record review

Exclusion Criteria:

* Patients enrolled in another interventional clinical trial
* An injured skin area for reinnervation at the volar side of the forearm, as well as an injured median or ulnar nerve.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with upper limb amputation (planned as well as accident related) with treatment resistant (phantom-and-or neuroma) pain.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2022-05-18 (Actual); Primary Completion 2023-08-02 (Actual); Study Completion 2023-08-02 (Actual)

PRIMARY OUTCOMES:
effects in use and reinervation (begin of sensation, localisation of sensation on the hand..) | 01.09.2020 - 31.03.2022
  Describtion of the effect of the use and reactivation of existing nerves in connection with the TSR in the delvelopment of phantom pain

OTHER OUTCOMES:
Date of targeted sensory reinervation (TSR) | 01.09.2020 - 31.03.2022
  Date, surgery to reinervate the nerve was performed
Start date and type of Physiotherapy | 01.09.2020 - 31.03.2022
  Type of physiotherapy: ultrasound, vibrational therapy, exercise...
Time between amputation and surgery | 01.09.2020 - 31.03.2022
  days, months or years
Cause of injury or disease | 01.09.2020 - 31.03.2022
  for example: accident
presence of phantom pain -and neuroma pain | 01.09.2020 - 31.03.2022
  patient survey and scale
concomittant treatment post TSR | 01.09.2020 - 31.03.2022
  dosage, indication and active agent of medication will be documented

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Gardetto, Doz.Dr, Principal Investigator — Brixsana Private Clinic; Smekal Vinzenz, Dr., Principal Investigator — AUVA Hospital Klagenfurt, Department of Orthopaedics and Traumatology
Locations (2):
- AUVA Hospital Klagenfurt, Klagenfurt, Carinthia, Austria
- Brixsana Private Clinic Center for Plastic, Aesthetic and Reconstructive Surgery with Hand Surgery Competence Center for Bionic Prosthetics, Brixen, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gardetto A, Baur EM, Prahm C, Smekal V, Jeschke J, Peternell G, Pedrini MT, Kolbenschlag J. Reduction of Phantom Limb Pain and Improved Proprioception through a TSR-Based Surgical Technique: A Case Series of Four Patients with Lower Limb Amputation. J Clin Med. 2021 Sep 6;10(17):4029. doi: 10.3390/jcm10174029. PMID 34501477